CLINICAL TRIAL: NCT01598103
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Cross-over Study to Evaluate the Efficacy, Safety and Tolerability of SAF312 in Subjects With Neurogenic Detrusor Overactivity Due to Spinal Cord Lesions Who Are Inadequately Managed by Antimuscarinic Therapy
Brief Title: Safety and Efficacy of SAF312 in Patients With Neurogenic Detrusor Overactivity Due to Spinal Cord Lesions
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSAF312A2202; 2010-021137-32 (EudraCT Number)
Record Dates: First submitted 2012-02-17; First posted 2012-05-15 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-04

CONDITIONS: Neurogenic Urinary Bladder; Neurogenic Bladder Disorder; Neurogenic Dysfunction of the Urinary Bladder; Neurogenic Bladder, Uninhibited; Neurogenic Bladder, Spastic
Keywords: Neurogenic detrusor overactivity; spinal cord lesions; spinal cord injury
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo to SAF312 (Placebo Comparator)
  Interventions: Drug: Placebo to SAF312
- SAF312 (Experimental)
  Interventions: Drug: SAF312

INTERVENTIONS:
Drug: SAF312 — One week of treatment in a BID (two times a day) regimen (hard gelatin capsules for oral use)
  Arms: SAF312
Drug: Placebo to SAF312 — One week of treatment in a BID (two times a day) regimen (hard gelatin capsules for oral use)
  Arms: Placebo to SAF312

SUMMARY:
This study will assess the safety, tolerability and efficacy of SAF312 in patients with overactive bladder disease due to spinal cord lesions. The overactive bladder of patients who qualify for this study is insufficiently managed by antimuscarinic therapy, or patients poorly tolerate the treatment with antimuscarinic drugs. The efficacy of SAF312 will be primarily determined via urodynamic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neurogenic detrusor overactivity due to spinal cord lesions
* Patients are inadequately managed by antimuscarinic medication and present with a cystometric bladder capacity of max. 400 mL

Exclusion Criteria:

* Chronic inflammation such as interstitial cystitis, bladder stones, hematuria of unknown origin, previous pelvic radiation therapy or previous or current malignant disease of the pelvic organs
* Pelvic or genitourinary tract anomalies including surgery or bladder disease other than detrusor overactivity impacting on bladder function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Maximum cystometric capacity (MCC) | 1 week
  Examined during filling cystometry as measured by changes from baseline following treatment for one week.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | 1 week
  Safety (physical exam, vital signs, haematology, coagulation parameters, clinical chemistry and urinalysis, ECG, pregnancy test, hand immersion test and PK [concentrations of SAF312 in blood]).
Bladder threshold vol, threshold pressure, instilled vol at first leak, detrusor pressure at first leak, vol/detrusor pressure at first sensation and at first desire to void, maximum detrusor pressure during filling/storage, bladder wall compliance | 1 week
  All parameters examined during filling cystometry as measured by changes from baseline following treatment for one week
Micturition or catheterization frequency | 1 week
  Changes from baseline, as measured by daily diaries.
Incontinence episodes | 1 week
  Changes from baseline as measured by daily diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, Murnau am Staffelsee, Germany
- Novartis Investigative Site, Nijmegen, Netherlands
- Novartis Investigative Site, Zurich, Switzerland

REFERENCES:
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Schafer W, Abrams P, Liao L, Mattiasson A, Pesce F, Spangberg A, Sterling AM, Zinner NR, van Kerrebroeck P; International Continence Society. Good urodynamic practices: uroflowmetry, filling cystometry, and pressure-flow studies. Neurourol Urodyn. 2002;21(3):261-74. doi: 10.1002/nau.10066. PMID 11948720
- [Background] Stohrer M, Blok B, Castro-Diaz D, Chartier-Kastler E, Del Popolo G, Kramer G, Pannek J, Radziszewski P, Wyndaele JJ. EAU guidelines on neurogenic lower urinary tract dysfunction. Eur Urol. 2009 Jul;56(1):81-8. doi: 10.1016/j.eururo.2009.04.028. Epub 2009 Apr 21. PMID 19403235
- See also: Results for CSAF312A2202 on the Novartis clinical trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=9783